CLINICAL TRIAL: NCT05663034
Title: CoMBat Insomnia: A Randomized Controlled Trial of Cognitive-Behavioral vs. Mindfulness-Based Treatment for TBI-Related Insomnia and Post-Traumatic Stress Symptoms
Brief Title: CBT-I vs. MBTI for Traumatic Brain Injury (TBI)-Related Insomnia and Post-Traumatic Stress Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Department of Defense Congressionally Directed Medical Research Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00356930; 141686 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Program)
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury; Insomnia; Depression; Post-traumatic Stress; Sleep; Memory Impairment; Cognitive Behavioral Therapy; Concussion, Brain; Head Injury; Brain Injury Traumatic Mild
Keywords: Traumatic Brain Injury; Insomnia; Posttraumatic Stress Symptoms; Depression; Concussion; Head Injury; Brain Injury; Cognitive Behavioral Therapy for Insomnia; Mindfulness-based Treatment for Insomnia
MeSH Terms: conditions — Brain Injuries, Traumatic; Sleep Initiation and Maintenance Disorders; Depression; Memory Disorders; Brain Concussion; Craniocerebral Trauma; Brain Injuries | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Prospective two-arm, single blind randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessment technicians will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy for insomnia (CBT-I) (Active Comparator): CBT-I treatment will involve a standardized 6-session blended intervention that combines cognitive and behavioral techniques. The core components include (1) education about sleep and insomnia, stimulus control (SC) and sleep restriction (SRT) (week 1); (2) sleep hygiene education (week 2); and (3) relaxation training, cognitive restructuring (to counter-arousal and address sleep-interfering cognitions), adherence monitoring, and adjusting the recommended sleep-wake schedule (weeks 3 through 6). The final session will also include a review of treatment content and relapse prevention. Common to all sessions is an initial review of participant diary data, charting progress, setting measurable goals, discussing adherence, and reinforcing learned skills.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBT-I)
- Mindfulness-based treatment for insomnia (MBTI) (Active Comparator): MBTI treatment will involve a standardized 6-session intervention which integrates the mindfulness training and exercises from mindfulness-based stress reduction (MBSR) with behavioral strategies based on sleep restriction therapy and stimulus control delivered within the context of mindfulness principles. Mindfulness principles include: 1) increase awareness of the mental and physical states that promote sleep (i.e., sleepiness), 2) shift sleep-related metacognitions to reduce hyperarousal, and 3) promote a mindful stance to respond when symptoms of insomnia arise. An overview of the treatment program, sleep education, and an introduction to the principles of mindfulness meditation is given (week 1). Then a combination of mindfulness meditations, sleep restriction, and stimulus control is conducted (week 2-6).
  Interventions: Behavioral: Mindfulness-based treatment for insomnia (MBTI)

INTERVENTIONS:
Behavioral: Mindfulness-based treatment for insomnia (MBTI) — A 6-week intervention that uses the principles and practices of mindfulness meditation along with behavioral strategies (stimulus control, sleep restriction therapy) to reduce symptoms of insomnia
  Arms: Mindfulness-based treatment for insomnia (MBTI)
Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) — Standard of care for adults with chronic insomnia. 6-week program that uses behavioral techniques to decrease psychophysiological arousal and increase sleep propensity to deepen and consolidate sleep.
  Arms: Cognitive behavioral therapy for insomnia (CBT-I)

SUMMARY:
This study is a prospective two-arm, single blind randomized controlled trial design to compare the clinical effectiveness of telemedicine-delivered, 6-session, standardized cognitive behavioral therapy for insomnia (CBT-I) and mindfulness-based treatment for insomnia (MBTI) in treating insomnia symptoms and ameliorating depressive symptoms in persons with mild to moderate TBI and comorbid Post-Traumatic Stress Symptoms (PTSS) and insomnia symptoms in a 360 patients. Participants will undergo assessment (psychosocial questionnaires, neurocognitive testing, sleep monitoring) at baseline, at the end of treatment, and at 2-, 6- and 12-weeks post-treatment. The primary outcome is sleep as measured by the Insomnia Severity Index (ISI).

DETAILED DESCRIPTION:
This study is a prospective two-arm, randomized single blind controlled trial design to compare the clinical effectiveness of telemedicine-delivered cognitive behavioral therapy for insomnia (CBT-I) and mindfulness-based treatment for insomnia (MBTI) in treating insomnia and ameliorating depressive symptoms in persons with mild to moderate TBI and comorbid symptoms of posttraumatic stress and insomnia. A cohort of n=360 adults with mild to moderate TBI and comorbid symptoms of posttraumatic stress and insomnia will be randomized to receive either telemedicine-delivered CBT-I or MBTI. Consistent with previous scientific literature, the interventions will be standardized and six sessions in length. All participants will wear an actigraph wrist monitor throughout the course of the project. All participants will also complete electronic sleep diaries throughout the course of the project. Participants will undergo assessment (psychosocial questionnaires, neurocognitive testing, sleep diaries, actigraphy, ambulatory EEG sleep monitoring) at baseline, at the end of treatment, and at 2-, 6- and 12-weeks post-treatment (12- and 24-weeks post randomization, respectively). The primary outcome is insomnia severity (ISI) and secondary outcomes are pre-sleep arousal, and depressive symptoms (PSAS; Patient Health Questionnaire (PHQ-8). Exploratory analyses will include neurocognitive functioning (ANAM) and pre-sleep arousal (PSAS).

ELIGIBILITY:
Inclusion Criteria:

1. Current or former member of the uniform services
2. Meet the Veterans Affairs Medical Center (VAMC) Department of Defense (DoD) criteria for TBI;
3. Time duration since traumatic brain injury (TBI) injury >90 days
4. Insomnia symptom duration >90 days
5. Endorse insomnia symptoms (Insomnia Severity Index [ISI] score > 10)
6. Display sufficient cognitive capacity to provide informed consent (Montreal Cognitive Assessment (MoCA) Z-score > -2)
7. >18 years of age
8. Access to and ability and to use computer.

Exclusion Criteria:

1. History of neurological diseases other than TBI and not attributable to TBI
2. Sleep apnea [apnea hypopnea index (AHI) >15; individuals with mild apnea (AHI > 5 and <15) will be informed, but allowed to participate]. Participants who use a continuous positive airway pressure (CPAP) device for sleep apnea will be eligible for participation if they are below the apnea/hypopnea cutoff while using CPAP, are adherent to using the device (> 4 hours/night 21/30 consecutive days) and agree to continue using the device during study participation.
3. Lastly, people using psychotropic medications may be included if they are on a stable dosage for the last three weeks prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia severity as assessed by the insomnia severity index (ISI) | At the end of treatment, and 2-, 6- and 12-weeks post treatment
  Insomnia symptoms and severity measured by insomnia severity index (ISI); score range: 0-28; Higher scores are associated with greater insomnia symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Luis Buenaver, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (5):
- United States (5):
  - Intrepid Spirit Center - Eglin Air Force Base, Eglin Air Force Base, Florida
  - Naval School Explosive Ordance Disposal - Eglin Air Force Base, Eglin Air Force Base, Florida
  - Walter Reed National Medical Military Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Madigan Army Medical Center, Fort Lewis, Washington